CLINICAL TRIAL: NCT02055508
Title: Physical Exercise Program in Lung Cancer Patients With Non-operable Disease Undergoing Palliative Treatment
Brief Title: POSITIVE - Study (Part III) Heidelberg
Acronym: POSITIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: National Center for Tumor Diseases, Heidelberg (Other); University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: POSITIVE-III-S-326/2013
Record Dates: First submitted 2013-12-12; First posted 2014-02-05 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Advanced NSCLC; First Line Treatment
Keywords: Exercise; Physical Activity; Palliative Care; Lung Cancer; NSCLC
MeSH Terms: conditions — Motor Activity; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Intervention Program (EIP) (Experimental): Inpatient periods: The combined resistance and endurance program consist of free weight and rubber band training for major upper and lower body muscle groups respectively of cycling/walking on an ergometer/treadmill 3x/week.
  Outpatient periods (3x/week at least two/one supervised training sessions): Supervised training sessions in the local outpatient training center will comprise of resistance exercise on machines and endurance training on an ergometer/treadmill. For non-supervised training session during the outpatient period participants will receive an exercise manual for individualized home-based exercising.
  In weekly phone calls, the advanced practice nurse will review adherence to the intervention and identify problems. Furthermore, the patients will also be asked the same questions as in the CMPC group.
  Interventions: Behavioral: Exercise Intervention; Other: Care-Management-Phone-Calls
- Care-Management-Phone-Calls (CMPC) (Active Comparator): Patients in this arm will receive a weekly "care-management-phone-call" (CMPC), performed by an advanced practice nurse (APN). The CMPCs are based on a structured questionnaire, reflecting pain, shortness of breath, disturbed sleep, exhaustion and distress and potentially treatment related side effects (e.g. infections, polyneuropathy, etc.). In case of demanding management of symptoms or complaints (e.g. uncontrolled pain or breathlessness) the treating physician is contacted by the APN to facilitate improvement.
  Interventions: Other: Care-Management-Phone-Calls

INTERVENTIONS:
Behavioral: Exercise Intervention
  Arms: Exercise Intervention Program (EIP)
Other: Care-Management-Phone-Calls

SUMMARY:
The investigators plan to evaluate, in a randomized, controlled phase III trial in patients with advanced non-small cell lung cancer (NSCLC), the effects of a 24-week exercise intervention program (EIP) on quality of life, physical functioning and immune function parameters. Eligible patients (n=250) will be enrolled in the Clinic for Thoracic Diseases, Heidelberg, over a time period of two years and followed up for a total of 12 months.

Patients will be randomized either to EIP plus Care Management Phone Calls (CMPC) versus CMPC alone (besides a proper symptom and side effect management CMPC ensures the potential influence of social contacts that can be anticipated for the patients in the intervention group).

Our primary aims are to investigate whether a combination of a partly supervised (in- and outpatient) and partly home-based endurance and resistance training improves quality of life (QoL) and lowers levels of fatigue (evaluation via the standardized and validated questionnaires FACT-L and MFI). In addition we propose to evaluate the effects of EIP on tumor specific immune responses. Biomarkers of immune function will be measured by cellular immunity and cytokine and chemokine panels.

Further secondary outcomes include measurement of anxiety, depression and demoralization, physical performance parameters (e.g. improvement in walk distance, muscle strength), as well as overall and progression free survival analyses.

The study builds on a previous feasibility study of a 8 weeks exercise intervention trial in patients with advanced NSCLC with the results being utilized in the design of the here proposed trial.

The investigators hypothesize that patients randomized in the exercise intervention group will show improved QoL and reduced fatigue, as well as improved physical functioning and increased tumor specific immune responses.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC stage IIIB/IV
* receiving systemic treatment (palliative radiotherapy accepted)
* BMI > 18
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2
* signed informed consent

Exclusion Criteria:

* serious active infection (i.e. requiring an iv antibiotic, antifungal or antiviral agent)
* inability to walk
* immobility (more than two days)
* previously untreated (non-irradiated or non-resected) symptomatic brain metastases;permitted are: (1) previously treated brain metastases [radiotherapy, surgery, dexamethasone dosage 8 mg per day, anti-epileptic therapy]; (2) asymptomatic brain metastases without additional therapy requirement
* severe neurologic impairment (e.g. apoplectic insult, Morbus Parkinson, pareses of extremities)
* severe cardiac impairment (e.g. cardiac insufficiency NYHA (New York Heart Association) > III, myocardial infarction within the last three months, unexplained syncopal events, severe cardiac arrhythmias, high grade aortic stenosis)
* severe respiratory insufficiency
* uncontrolled pain
* abuse of alcohol or drugs reducing compliance to the study
* bone metastasis inducing skeletal fragility
* any circumstance that would impede ability to give informed consent or adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
QoL: Physical Well-Being (FACT-L) | assessed after 12 weeks of enrolement
  The FACT-L (Functional Assessment of Cancer Therapy-Lung) questionnaire comprises of 36 items and deter-mines the quality of life in patients with lung cancer. It is separated in the subcategories "physical well-being" (PRIMARY OUTCOME), "emotional well-being", "social well-being", "functional well-being and disease-specific items". It is widely used in clinical studies and was already applied in exercise intervention studies in lung cancer patients
General Fatigue (MFI) | assessed after 12 weeks of enrolement
  The MFI (Multidimensional Fatigue Inventory) questionnaire (20 items) evaluates the extent of chronic fatigue and is divided into the 5 subscales "general fatigue", "physical fatigue", "mental fatigue", "reduced motivation" and "reduced activity". The MFI questionnaire is widely used in oncological studies and an adequate number of comparative samples exists.

SECONDARY OUTCOMES:
Physical Performance (endurance and strength capacity) | assessed every 3 month after enrolement until month 12
  6-Minute Walk Test (endurance capacity) The 6 minute walk test is feasible and safe to determine patients physical capacity. Patients are instructed to walk in 6 min. as many meters as possible with oxygen saturation and pulse rate being measured concomitantly.
  Hand-held Dynamometry (isometric strength capacity) The hand-held dynamometry is a standardized instrument to measure muscular strength. In the study 6 major muscle groups of upper and lower extremities will be assessed for their isometric power.
Psychosocial Parameters (e.g. depression, anxiety, demoralization) | assessed every 3 month after enrolement until month 12
  PHQ(Ultra-Brief Patient Health Questionnaire)-4 :
  The PHQ-4 (Ultra-Brief Patient Health Questionnaire) questionnaire is a short instrument comprising of 4 items to detect the extent of depression and anxiety. It provides sufficient diagnostic accuracy for major depression and can be used as a screening instrument in cancer populations.
  DS (Demoralization Scale) The demoralization scale (DS) is a relatively new developed questionnaire to detect the extent of existential distress in cancer patients. The German version was validated in 2011 and comprises of 24 questions. The results of the validation showed that the concept of demoralization is a useful instrument to describe the different states of existential distress and the individual incapacity to cope effectively with stressful situations.
Overall survival | for the period of 1 year after enrolement
progression-free survival | for the period of 1 year after enrolement

OTHER OUTCOMES:
Adverse Events | baseline until 6 month after enrolement
  Safety analyses will be based on Adverse Events (AE´s), Severe Adverse Events (SAE´s), and Suspected Unexpected Serious Adverse Reaction (SUSARs) recorded during the study. Of particular interest are AEs, SAEs and SUSARs deemed to be potentially causally related to the endurance and resistance training.
Translational Program / Immunology | baseline, 3 & 6 month after enrolement
  Quantification (Q) of immune cells: Multicolor flow cytometry from cryopreserved Peripheral Blood Mononuclear Cell (PBMC), CD (cluster of differentiation) 4+ and CD 8+ T cells, effector, naïve and activated T cells, regulatory T cells (Treg) and their functional subsets, natural killer cells, B cells, monocytes and monocyte-derived myeloid suppressor cells will be assessed.
  Q. of tumor antigen reactive effector/memory T cells: Will be done by interferon gamma Enzyme Linked Immuno Spot Assays from PBMC using a panel of defined tumor antigens presented by generated autologous dendritic cells as antigen presenting cells and purified T cells as responder cells.
  Detection of tumor reactive Treg: Will be done by established Treg specificity assay based on the increased suppressive activity of specifically activated regulatory T cells.
  Q. of key immune effector molecules: Will be done for app. 14 different cytokines and chemokines from cryopreserved serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thomas, Prof. Dr., Principal Investigator — Thoracic Oncology Clinic for Thoracic Diseases/University of Heidelberg; Joachim Wiskemann, Dr., Principal Investigator — National Center for Tumor Diseases (NCT); Simone Hummler, Dr., Principal Investigator — Thoracic Oncology Clinic for Thoracic Diseases/University of Heidelberg
Locations (1):
- Thoracic Oncology Clinic for Thoracic Diseases, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Titz C, Hummler S, Schmidt ME, Thomas M, Steins M, Wiskemann J. Exercise behavior and physical fitness in patients with advanced lung cancer. Support Care Cancer. 2018 Aug;26(8):2725-2736. doi: 10.1007/s00520-018-4105-5. Epub 2018 Feb 26. PMID 29480444
- [Derived] Wiskemann J, Hummler S, Diepold C, Keil M, Abel U, Steindorf K, Beckhove P, Ulrich CM, Steins M, Thomas M. POSITIVE study: physical exercise program in non-operable lung cancer patients undergoing palliative treatment. BMC Cancer. 2016 Jul 19;16:499. doi: 10.1186/s12885-016-2561-1. PMID 27430336